CLINICAL TRIAL: NCT06117670
Title: Gamma-irradiated Amniotic Membrane Graft in Posterior Colporrhaphy. A Pilot One Arm Clinical Trial
Brief Title: Gamma-irradiated Amniotic Membrane Graft in Posterior Colporrhaphy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Mostafa, Dr, Ain Shams Maternity Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD81/2023
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Rectocele; Female; Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; sexual satisfaction; POP-Q
MeSH Terms: conditions — Rectocele; Pelvic Organ Prolapse; Orgasm

STUDY DESIGN:
Intervention Model Description: patients will undergo posterior colporrhaphy using gamma-irradiated amniotic membrane as a graft
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- amniotic membrane graft (Experimental): women with posterior vaginal prolapse will be enrolled and posterior colporrhaphy will be done with the application of sterilized (gamma irradiated) amniotic membrane as a graft.
  Interventions: Combination Product: posterior colporrhaphy using gamma-irradiated amniotic membrane as a graft

INTERVENTIONS:
Combination Product: posterior colporrhaphy using gamma-irradiated amniotic membrane as a graft — Posterior colporrhaphy with application of the gamma-irradiated amniotic membrane graft will be done

SUMMARY:
The goal of this clinical trial is to test the benefit of using gamma-irradiated amniotic membrane as a graft in surgical repair for women with posterior vaginal wall defects. The main question it aims to answer is:

• Is posterior colporrhaphy using gamma-irradiated amniotic membrane as a graft effective?

Participants will undergo posterior colporrhaphy, which will be modified by adding gamma-irradiated amniotic membrane as a graft during the repair.

DETAILED DESCRIPTION:
• Methodology:

1. Protocol approval will be sought from the research ethical committee.
2. Enrolment: The patients will be recruited from the outpatient gynecology clinic of Ain Shams University Maternity Hospital (ASUMH).
3. History, examination, and routine investigations will be done to identify eligible patients.

   History taking including (personal history, age, menopausal, medical history, and surgical history), as well as symptoms score using Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6) part of the Pelvic Floor Distress Inventory Short Form 20. Also, sexual function will be assessed by Female Sexual Function Index Questionnaire.

   Clinical examination: including (general examination, abdominal examination and pelvic examination and POP-Q.

   Routine investigations: complete blood count and other preoperative tests as needed.
4. Written informed consent will be sought from the patients after proper counseling.
5. Surgical procedure:

   Posterior colporrhaphy with application of the amniotic membrane graft will be done as follows:

   Steps of conventional posterior colporrhaphy:
   * A midline incision is extended from the perineal body to the vaginal apex or to the cephalad border of a small or distal rectocele.
   * The Denonvillier's fascia is mobilized from the vaginal epithelium, leaving as much of the tissue as possible attached laterally to the levator fascia.
   * Gamma irradiated Sterilized freeze-dried (lyophilized) amnion grafts will be obtained from the Egyptian Atomic Energy Authority and prepared according to the method of Antounians (2019). Multiple procedures are used to sterilize acellular amniotic membranes, the final of which being gamma irradiation. For tissue allograft sterilisation, gamma radiation is claimed to be the most reliable and successful method. Many tissue banks have employed it to sterilise tissues. The clinical function of the amniotic membrane is unaffected by gamma radiation 11. The most frequent dose for sterilising medical goods is 25 kilogram. This graft has the advantage of complete sterilization and is valid on shelf for 5 years as it is dried. Posterior vaginal wall amniotic membrane graft can be placed on the posterior vaginal wall, between the rectal fascia and the vagina, anchored distally at the uterosacral ligaments, and dorsally at the levator ani muscle. The excess amniotic membrane graft is trimmed off, usually around 1-2 cm on each side.
   * After obvious defects in the rectal muscularis are repaired, the fascia is plicated in the midline with interrupted or continuous sutures using vicryl 0 sutures.
   * When a defective perineal body or perineal membrane is present, reconstruction is performed after accompanying posterior colporrhaphy.
   * The superficial muscles of the perineum and bulbocavernous fascia are plicated in the midline and the skin closed as in an episiotomy repair using vicryl 2/0 sutures.
   * Detachments of the inferior portion of the Denonvillier's fascia from the perineal body are also corrected.

   Postoperative instructions and care:
   * Vaginal pack will be left as a compression and will be removed the following day.
   * Urinary catheter: will be left for 24hours then removed.
   * Postoperative clinical assessment by POP-Q.
   * Patients will be instructed to:
   * Mobilize to reduce risk of deep vein thrombosis.
   * Bath or shower as normal routine.
   * Avoid using tampons for 6 weeks.
   * Avoid sexual intercourse for at least 6weeks.
   * Avoid constipation; by drinking plenty of water and fluids, eating fruit and green vegetables, and any constant cough is to be treated promptly.
   * Avoid heavy lifting to reduce the risk of the prolapse recurrence.
6. Follow up schedule:

   Follow up of all patients will be done in both groups at 3 and 6 months (symptoms +/- examination as needed).
7. Data collection and recording. Data will be collected and recorded in case report form. Detection bias will be avoided by blinding the outcome assessor.
8. Statistical analysis will be done to get the results.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed as posterior vaginal wall prolapse: bulging of front wall of rectum into the vagina due to weakening of pelvic support system and thinning of rectovaginal septum.
* Women aged 30-60 years.
* BMI 20-35 kg/m2
* Planned for surgical correction

Exclusion Criteria:

* Patients with:
* Immuno-compromise e.g. Patients receiving chemotherapy, steroids.
* Severe anaemia (Hb<10)
* conditions that require concomitant reconstructive pelvic floor surgery e.g., anterior and/or apical compartment prolapse.
* Conditions that lead to increase intra-abdominal pressure e.g.,chronic obstructive pulmonary disease.
* Uncontrolled medical disorders (diabetes, hypertension, asthma).

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
POP-Q | first week postoperative
  Prolapse assessment using the prolapse quantification system of the International Continence Society (POP-Q)
POPDI-6 score | at 3 months, and at 6 months postoperative
  Assessment of symptoms score using Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6) part of the Pelvic Floor Distress Inventory Short Form 20. Scale from 0 to 100, the higher score indicates worse condition.

SECONDARY OUTCOMES:
sexual satisfaction | at 3 months, and at 6 months postoperative
  to measure sexual satisfaction using female sexual function index questionnaire The Female Sexual Function Index (FSFI) was developed to assess six domains of female sexual function (sexual desire, sexual arousal, lubrication, orgasm, satisfaction, and pain).
  Items are scored on a five-point Likert scale with low scores indicating lower levels of sexual functioning. Fifteen items also include a zero score as a sixth response option indicating no sexual activity in the past 4 weeks.
  Range: 2 to 36.
wound complications | within 6 months postoperative
  Wound infection or wound dehiscence as detected clinically and /or CRP and vaginal swab as needed
Intraoperative complications | Intraoperative
  occurrence of intraoperative bladder or bowel injury

CONTACTS AND LOCATIONS:
Overall Officials: Ihab FS Eldin Allam, MD, Study Chair — Ain Shams University; Ahmed M Abbas, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the results, and the analytic code after publication of the study manuscript after the study has completed
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available after publication, for 10years.
Access Criteria: data will be sent via e-mail upon reasonable request (raneyah@med.asu.edu.eg)